CLINICAL TRIAL: NCT01830530
Title: HIGH Altitude CArdiovascular REsearch in the ANDES
Acronym: HIGHCARE-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09F102
Record Dates: First submitted 2013-02-18; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-02

CONDITIONS: Hypertension; High Altitude
Keywords: arterial hypertension; high altitude; hypobaric hypoxia; combination treatment; angiotensin receptor blocker; calcium antagonist
MeSH Terms: conditions — Hypertension; Altitude Sickness | interventions — Telmisartan; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telmisartan/nifedipine (Experimental): Subjects treated with telmisartan 80 mg (1 capsule daily in the morning) plus nifedipine slow release 30 mg (1 capsule daily in the morning) combination
  Interventions: Drug: Telmisartan; Drug: Nifedipine
- Placebo (Placebo Comparator): Two tablets containing placebo daily in the morning
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Telmisartan — Subjects treated with telmisartan 80 mg (1 capsule daily in the morning) plus nifedipine slow release 30 mg (1 capsule daily in the morning) combination
  Other Names: Pritor; Micardis
  Arms: Telmisartan/nifedipine
Drug: Nifedipine — Subjects treated with telmisartan 80 mg (1 capsule daily in the morning) plus nifedipine slow release 30 mg (1 capsule daily in the morning) combination
  Other Names: Adalat
  Arms: Telmisartan/nifedipine
Drug: placebo — two tablets daily in the morning
  Arms: Placebo

SUMMARY:
This study is aimed to assess the efficacy of combined treatment with two antihypertensive agents (telmisartan and nifedipine) in subjects with mild hypertension exposed to high altitude.

DETAILED DESCRIPTION:
This is a parallel group, prospective, double-blind, placebo controlled randomized trial, comparing the effects of combination of two antihypertensive agents (telmisartan/nifedipine)with placebo in hypertensive subjects exposed to high altitude. The principal objectives are:

1. to assess the response of BP to high altitude exposure in hypertensive subjects residing at sea level
2. To assess the efficacy and safety of combination of telmisartan 80 mg with nifedipine GITS 30 mg in preventing a possible excessive BP increase in hypertensive subjects exposed to high altitude.

The following data will be collected during the study at the different steps:

* Clinical history
* Symptoms and adverse events questionnaire
* Conventional BP and heart rate (HR) measurement - seated measurements with a validated oscillometric device will be performed after at least 5 minutes rest on non-dominant arm; two measurements will be performed 1-2 minutes apart and their average will be used in the analyses
* Vital signs:

respiratory rate - will be measured manually over 60 seconds body height and weight, waist circumference blood oxygen saturation (SpO2)

* Lake Louise Score
* 24 h ambulatory blood pressure monitoring (ABPM; AND TM2430, AND, Japan)
* Echocardiography
* Arterial properties assessment
* Six minute walking test (6MWT)
* Cardiopulmonary Exercise Test (CPET) in a subgroup of subjects
* Polysomnography with a portable device
* Pulmonary function tests (only at sea level baseline visit)
* Fluid balance chart
* Blood and urine analyses: Visit 1: electrolytes, creatinine, estimated glomerular filtration rate (eGFR), glycemia, renin, angiotensin, aldosterone, plasma catecholamines, 24 h urinary sodium excretion, carbonic anhydrase activity and isoenzyme expression (in 50 randomly selected subjects), samples for genetic studies. Visit 2: electrolytes, creatinine, eGFR. Visit 3: complete blood count, electrolytes, creatinine, eGFR, glycemia, insulin, renin, angiotensin, aldosterone, plasma catecholamines, classic urinalysis, microalbuminuria, 24 h urinary sodium excretion, carbonic anhydrase activity and isoenzyme expression (in 50 subjects selected at Visit 1). Visit 4: electrolytes, creatinine, eGFR, glycemia, insulin, renin, angiotensin, aldosterone, plasma catecholamines, 24 h urinary sodium excretion, carbonic anhydrase activity and isoenzyme expression (in 50 subjects selected at Visit 1)

ELIGIBILITY:
Inclusion Criteria:

* Permanent residence at low (<500 m) altitude
* Conventional systolic BP (average of two measurements) 140-159 mmHg or conventional diastolic BP 90-99 mmHg in subjects untreated or after 4 weeks of washout
* Mean daytime systolic BP ≥135 and <150 mmHg and/or mean daytime diastolic BP ≥85 and <95 mmHg in subjects untreated or after 4 weeks of washout
* Written informed consent to participate in the study

Exclusion Criteria:

* Conventional systolic BP (average of two measurements) ≥150 mmHg and conventional diastolic BP ≥95 mmHg in treated subjects
* Regular use of two or more antihypertensive drugs (with the exception of subjects on two antihypertensive drugs in low doses)
* Treated antihypertensive subjects in whom withdrawal of treatment is deemed unethical by the investigator (e.g. because of the existence of compelling indications other than hypertension for continuous use of previously used antihypertensive agent)
* Contraindications (including a history of adverse reactions) to angiotensin receptor blockers or calcium antagonists
* History of serious mountain sickness
* Subjects who over 3 months preceding inclusion in the study spent considerable (> 1 week) amount of time at altitudes above 2500 m.
* Cardiovascular diseases other than hypertension (coronary heart disease, heart failure, atrial fibrillation, valvular or congenital heart disease, cardiomyopathies, cerebrovascular disease, peripheral artery disease, aortic aneurysm)
* Suspected or confirmed secondary hypertension
* Diabetes mellitus
* Serious respiratory disorders
* Other conditions deemed relevant by the investigator (including liver disease, renal disease, thyroid disorders)
* BMI ≥35 kg/m2
* Upper arm circumference >32 cm
* known severe obstructive sleep apnea (apnea-hypopnea index > 30 or use of CPAP) or excessive daytime sleepiness (Epworth Sleepiness Scale > 10)
* Pregnancy
* Premenopausal women not using effective contraceptive methods
* Elevated probability of noncompliance with the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Effect of study treatment on 24 h ambulatory systolic blood pressure at high altitude | After 6 weeks of study treatment, during high altitude visit
  Difference in 24 h ambulatory systolic BP at high altitude (Visit 4) between combination therapy group and placebo group

SECONDARY OUTCOMES:
Effect of study treatment on ambulatory blood pressure at high altitude (other variables) | After 6 weeks of study treatment, during high altitude visit
  Differences in other ambulatory blood pressure (BP) variables (including 24 h diastolic BP, daytime and night-time BP, nocturnal fall of BP) at high altitude (V4) between combination therapy and placebo groups
Lake Louise Score | After 6 weeks of study treatment, during high altitude visit
  Differences in Lake Louise Score (score of acute mountain sickness severity) between groups
Effect of high altitude on ambulatory blood pressure | After 6 weeks of study treatment, during high altitude visit
  Change in ambulatory blood pressure between sea level condition and high altitude in both treatment groups
Effect of high altitude on conventional blood pressure | After 6 weeks of study treatment, during high altitude visit
  Change in conventional blood pressure between sea level condition and high altitude in both groups
Effect of study treatment on conventional blood pressure at high altitude. | After 6 weeks of study treatment, during high altitude visit
  Difference in conventional systolic and diastolic blood pressure at high altitude (Visit 4) between combination therapy group and placebo group
Rate of adverse events | After 6 weeks of treatment plus up to 1 additional week of treatment needed for high altitude visit (study end).
  Differences in rate of adverse events between groups.
Effect of study treatment on ambulatory heart rate at high altitude | After 6 weeks of study treatment, during high altitude visit
  Differences in ambulatory heart rate (HR) variables (including 24 h, daytime and night-time HR, and nocturnal fall of HR) at high altitude (V4) between combination therapy and placebo groups

OTHER OUTCOMES:
Differences in other variables assessed in the study at high altitude between treatment groups | high altitude visit ( Visit 4)
  Differences between treatment groups in polysomnographic data, arterial stiffness, blood tests, echocardiography data assessed at high altitude
blood pressure response at sea level | Sea level visit (3) and high altitude visit (4)
  Changes in polysomnographic data, arterial stiffness, blood tests, echocardiography data between sea level condition and high altitude

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, PhD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

REFERENCES:
- [Derived] Caravita S, Faini A, Baratto C, Bilo G, Macarlupu JL, Lang M, Revera M, Lombardi C, Villafuerte FC, Agostoni P, Parati G. Upward Shift and Steepening of the Blood Pressure Response to Exercise in Hypertensive Subjects at High Altitude. J Am Heart Assoc. 2018 Jun 9;7(12):e008506. doi: 10.1161/JAHA.117.008506. PMID 29886423
- [Derived] Bilo G, Villafuerte FC, Faini A, Anza-Ramirez C, Revera M, Giuliano A, Caravita S, Gregorini F, Lombardi C, Salvioni E, Macarlupu JL, Ossoli D, Landaveri L, Lang M, Agostoni P, Sosa JM, Mancia G, Parati G. Ambulatory blood pressure in untreated and treated hypertensive patients at high altitude: the High Altitude Cardiovascular Research-Andes study. Hypertension. 2015 Jun;65(6):1266-72. doi: 10.1161/HYPERTENSIONAHA.114.05003. Epub 2015 Apr 20. PMID 25895588